CLINICAL TRIAL: NCT03465358
Title: Validation of Completion of Items 18, 19 and 22 of the Motor Function Measure (MFM) on a Digital Tablet
Acronym: MFM-tablet
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0851
Record Dates: First submitted 2018-03-08; First posted 2018-03-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Neuromuscular Diseases
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Items completion — Patients will complete his Motor Function Measure in the usual way, except items 18, 19 and 22 which will be completed twice: once using conventional material and once on a digital tablet.
  The order of completion between conventional material or digital tablet will be allocate randomly.

SUMMARY:
Motor Function Measure (MFM) is a validated tool assessing the motor function of neuromuscular patients constituted of 32 items. Despite standardized Motor Function Measure (MFM) training sessions, there is still an inter-individual variability in the items' scoring procedure, depending for example on the subjectivity of the therapist.

Among the 32 items of the MFM, 3 currently require the use of a paper, and could be automated by using a digital tablet. It is the item 18 where the patient traces the edge of a Compact Disc, item 19 requiring to draw loops inside a frame and item 22 requiring to place a finger on each standardized cases. The reproducibility of these 3 items could be improved with the use of a digital tablet and the development of a software allowing to computerize the scoring procedure. The second interest is to implement directly the MFM data in the MFM base.

The hypothesis is that the difference of scoring of these 3 items between digital tablet versus paper completion is enough low to use indifferently each completion in patients with a neuromuscular disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a labelled neuromuscular disease
* Patients with Motor Function Measure in one of the participating services during their usual follow-up
* Patients who received the information and did not object to participating in the study or their parents for the children

Exclusion Criteria:

* Patients passing their Motor Function Measure as part of another research protocol

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with neuromuscular disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
Comparison scoring between items completed using conventional material or on a digital tablet. | 1 day
  The comparison of scores between usual test (paper) versus digital tablet test, for the item 18, 19 and 22 of the Motor Function Measure.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Service de Rééducation Fonctionnelle Pédiatrique - L'Escale (Aile A1) - Hôpital Femme Mère Enfant - GHE, Bron
  - Centre de référence MNM Adulte Grenoble Consultation Maladies Neuromusculaires Adultes - CHU Michallon, Grenoble
  - Centre de référence MNM adulte Lyon Hôpital de la Croix Rousse Bâtiment P, Lyon
  - Service de Médecine Physique et de Réadaptation Pédiatrique Hôpital de Bellevue, CHU, Saint-Etienne
  - Centre de référence MNM Adulte Saint Etienne CHU Hôpital Nord-service neurologie, Saint-Priest-en-Jarez

IPD SHARING:
Plan to Share IPD: No